CLINICAL TRIAL: NCT07126756
Title: Visual Outcomes Comparison of LASIK Using Wavefront Optimized and SMILE
Brief Title: LASIK iDesign vs SMILE
Acronym: TG-LASIK vs SM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Collaborators: United States Army Aeromedical Research Laboratory (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2024.066
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: Prospective randomized contralateral study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LASIK using iDesign (Active Comparator): LASIK guided by iDesign
  Interventions: Device: STAR S4 IR Excimer Laser System
- SMILE (Experimental): SMILE Refractive Surgery
  Interventions: Device: VisuMax 400 Surgical Laser

INTERVENTIONS:
Device: STAR S4 IR Excimer Laser System — LASIK with iDesign
  Other Names: iDesign Refractive Studio
  Arms: LASIK using iDesign
Device: VisuMax 400 Surgical Laser — small incision lenticule extraction technique
  Arms: SMILE

SUMMARY:
The study will compare the 6-month visual outcomes (i.e., visual acuity, contract sensitivity, higher order aberrations), quality of vision (i.e., double vision, glare, starburst, halos, etc.) and dry eye symptoms of patients undergoing contralateral LASIK using iDesign and SMILE surgery.

DETAILED DESCRIPTION:
Both SMILE and LASIK treatments are FDA-approved and are both performed routinely as standard of care surgery in the US Military. However, there is limited literature comparing quality of vision after LASIK using iDesign and SMILE refractive surgery. Our objective is to study the 6-month visual outcomes (high and 5% low contrast visual acuity, refractive error, higher order aberrations) and subject reported quality of vision (i.e., double vision, glare, starburst, halos, etc.) and dry eye symptoms using the PROWL and SPEED questionnaires following contralateral LASIK using iDesign and SMILE surgery. This is a prospective randomized contralateral study, including 57 subjects. Once consented to participate in the study, subjects will have a comprehensive ocular examination to determine eligibility to undergo simultaneous SMILE surgery in one eye and LASIK using iDesign on the contralateral eye to correct myopia. Surgical treatment will be randomized so there is a 50% chance to receive SMILE on the right eye and LASIK on the contralateral eye. Subjects will receive standard of care topical ophthalmic antibiotic and steroid drops. Visual outcomes and patient self-reported symptoms will be assessed at day 1, week 2, month 1, month 3, and month 6.

ELIGIBILITY:
Inclusion Criteria:

1. Nearsightedness (myopia) between -2.00 diopters and -8.00 diopters
2. Have similar levels of nearsightedness in each eye (2D or less difference between eyes)
3. Less than or equal to 3.00 diopters of astigmatism
4. Total spherical equivalent (SE) of no more than -8.0 D
5. Tricare Prime/Select Beneficiary (military health insurance)
6. Residing within 60 miles radius from Lackland AFB

Exclusion Criteria:

1. Subjects with corneal abnormal findings including signs of keratoconus, keratoconus suspect, abnormal corneal topography, epithelial basement membrane disease, pellucid marginal degeneration, corneal degenerations, progressive and unstable myopia, irregular or unstable corneal mires on central keratometry images, and volunteers whose corneal thickness would cause anticipated treatment would violate the posterior 250 microns (um) of corneal stroma from the corneal endothelium.
2. Subjects with active collagen vascular, connective tissue, autoimmune or immunodeficiency diseases
3. Pregnant or nursing females (pregnancy test will be performed on females subjects of childbearing potential)
4. Systemic disease likely to affect wound healing, such as uncontrolled diabetes and severe atopy
5. Any ocular disease such as advanced/uncontrolled glaucoma, severe dry eye, active eye infection or inflammation, recent herpes eye infection or problems resulting from past infection.
6. 0.25 or 0.50 of manifest astigmatism in the eye randomized to SMILE
7. Taking the medication Isotretinoin (Accutane) or antimetabolites for any medical condition.
8. Potential candidate who cannot provide Informed Consent will not be allowed to participate.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Eyes With Uncorrected Visual Acuity of 20/16 or Better at 6-month Post-Op | 6-month Post-Op
  Post-operative uncorrected visual acuity of 20/16 or better measure using the ETDRS chart reported as percentage of subjects; unit = percentage eyes with Uncorrected Visual Acuity

SECONDARY OUTCOMES:
Difference in High Contrast Visual Acuity at 6-month Post-Op | 6-month Post-Op
  Mean uncorrected high contrast visual acuity measure using the ETDRS chart measure at 6-month Post-Op; unit = LogMAR
Difference in residual Refractive Error at 6-month Post-Op | 6-month Post-Op
  Residual mean refractive error measure with phoropter at 6-month Post-Op; unit = Diopters (D)
Difference in Low Contrast Visual Acuity at 6-month Post-Op | 6-month Post-Op
  Mean uncorrected low contrast visual acuity measure using the 5% ETDRS chart measure at 6-month Post-Op; unit = LogMAR
Difference in residual Higher Order Aberrations at 6-month Post-Op | 6-month Post-Op
  Mean Higher Order Aberrations measure by iDesign 2.0 Refractive Studio at 6-month Post-Op; unit = root mean square
Difference in overall satisfaction questionnaire score at 6-month Post-Op | 6-month Post-Op
  Mean Subject Satisfaction Score with the surgery outcome using the Patient-Reported Outcomes with LASIK Symptoms and Satisfaction (PROWL-SS) Questionnaire at 6-month Post-Op. The score ranges from 1 (completely satisfied) to 6 (completely dissatisfied). Lower value indicates higher satisfaction.
Difference in overall Dry Eye questionnaire score at 6-month Post-Op | 6-month Post-Op
  Mean Standard Patient Evaluation of Eye Dryness (SPEED) Questionnaire score at 6-month Post-Op. Possible dry eye symptoms score ranges from 0 (never) to 3 (Constant). Higher value indicates worse dry eye symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Charisma B Evangelista, MD, Principal Investigator — Joint Warfighter Refractive Surgery Center, Wilford Hall Ambulatory Surgical Center
Locations (1):
- Joint Warfighter Refractive Surgery Center, Wilford Hall Ambulatory Surgical Center, Lackland Air Force Base, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma KK, Manche EE. Patient-reported quality of vision in a prospective randomized contralateral-eye trial comparing LASIK and small-incision lenticule extraction. J Cataract Refract Surg. 2023 Apr 1;49(4):348-353. doi: 10.1097/j.jcrs.0000000000001127. PMID 36539217
- [Background] Bharti S, Bains HS. Active cyclotorsion error correction during LASIK for myopia and myopic astigmatism with the NIDEK EC-5000 CX III laser. J Refract Surg. 2007 Nov;23(9 Suppl):S1041-5. doi: 10.3928/1081-597X-20071102-11. PMID 18047004